CLINICAL TRIAL: NCT00766181
Title: An Evaluation of Parent and Nurse Satisfaction Associated With Pediatric Peripheral Intravenous Catheter Placement Using Standard of Care vs. ZingoTM in the Emergency Department
Brief Title: Satisfaction With Pediatric Intravenous Catheter Placement in the Emergency Department
Status: Terminated | Type: Observational
Why Stopped: Product withdrawn from distribution
Sponsor: Anesiva, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Mitra Sadeghi, Pharm.D., Anesiva, Inc.
Other Study IDs: 113-03P
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2008-11

CONDITIONS: Intravenous Placement Procedure
Keywords: IV placement; Parent satisfaction level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Lifestyle: Observatonal
- 2: Lifestyle: Observational
  Interventions: Behavioral: Zingo TM (lidocaine hydrochloride monohydrate) powder intradermal injection system

INTERVENTIONS:
Behavioral: Zingo TM (lidocaine hydrochloride monohydrate) powder intradermal injection system — 0.5 mg lidocaine hydrochloride
  Groups: 2: Lifestyle

SUMMARY:
The purpose of this study is to determine the satisfaction among parents and nurses of pediatric patients with IV catheter placement in the Emergency Department.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate whether the proportion of parents satisfied with their child's IV placement procedure is higher after the introduction of Zingo compared to standard of care and to evaluate changes in nursing staff satisfaction with performing IV placement procedures after using Zingo prior to IV placement compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* PHASE A: Parent of a pediatric patient from the age of 3 to 18 years of age who requires a peripheral IV placement in the Emergency Department
* Parent must be able to read and understand English and provide written informed consent
* Parent must be present during the IV placement
* PHASE B: Parent did not participate in Phase A
* Nurse has completed Zingo TM in-service training prior to participation
* Zingo is used prior to performing the IV placement procedure

Exclusion Criteria:

- Parent of patient with a serious unstable medical or psychological condition that would compromise participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pediatric patients in Emergency Department requiring peripheral IV catheter placement.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-02 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Parent's satisfaction with IV placement procedure | 18 weeks

SECONDARY OUTCOMES:
Nurse'e satisfaction with performing IV placement | 18 weeks

REFERENCES:
- See also: Anesiva home page — http://www.anesiva.com/
- See also: Zingo Product Information — http://www.zingo.com